CLINICAL TRIAL: NCT05945550
Title: Comparison of Complication Rates Between Initial and Re-operative Anterior Lumbar Interbody Fusion Surgery: Is There a Difference?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 038.SUR.2020.A
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Lumbar Spondylolisthesis; Lumbar Spine Degeneration
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify the current mortality rate for initial ALIF procedures. Establish/prove mortality rates for this operation have dropped in the past decade.

DETAILED DESCRIPTION:
Establish the mortality rate for "re-do" ALIF procedures [i.e., is it different than that of initial ALIF procedures and - if so - postulate that there are interventions that can be done in the pre-operative period to ameliorate that risk. This study is not designed to "prove" the latter hypothesis.]

This is a single sample study where medical records will be searched by CPT codes for ALIF codes (e.g. 22558, 22585, 22845, etc.) by trained researcher(s) at participating Methodist facilities going back 5-10 years to see if 1500-3500 cases can be identified within that time period.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 17 years of age, patients having had ALIF procedures as defined by CPT codes at participating Methodist facilities during 2010-2020 targeted.

Exclusion Criteria:

* Pediatric patients (as defined by age <18 years old), pregnant women and incarcerated individuals. We do not anticipate any of these in an elective spine surgery group of patients. If they have emergency spine surgery it is normally not an ALIF.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 17 years of age, patients having had ALIF procedures as defined by CPT codes at participating Methodist facilities during 2010-2020 targeted.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2020-12-28 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Establish/prove mortality rates | 5 years
  Establish mortality rates of patients for this operation have dropped in the past decade.

SECONDARY OUTCOMES:
Establish the mortality rate for "re-do" ALIF procedures [ | 5 years
  Establish the patient's mortality rate, postulate that there are interventions that can be done in the pre-operative period to ameliorate that risk.

CONTACTS AND LOCATIONS:
Overall Officials: Reed Donald, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual.

REFERENCES:
- [Background] Weiss AJ, Elixhauser A. Trends in Operating Room Procedures in U.S. Hospitals, 2001-2011. 2014 Mar. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #171. Available from http://www.ncbi.nlm.nih.gov/books/NBK201926/ PMID 24851286
- [Background] 2. NA. (2019). Data on Spinal Fusion Surgery. Retrieved from HealthTrust: The Source Magazine: https://healthtrustpg.com/thesource/clinical-connection/data-on-spinal-fusion-surgery/
- [Background] Martin BI, Mirza SK, Spina N, Spiker WR, Lawrence B, Brodke DS. Trends in Lumbar Fusion Procedure Rates and Associated Hospital Costs for Degenerative Spinal Diseases in the United States, 2004 to 2015. Spine (Phila Pa 1976). 2019 Mar 1;44(5):369-376. doi: 10.1097/BRS.0000000000002822. PMID 30074971
- [Background] Neifert SN, Martini ML, Hanss K, Rothrock RJ, Gilligan J, Zimering J, Caridi JM, Oermann EK. Large Rises in Thoracolumbar Fusions by 2040: A Cause for Concern with an Increasingly Elderly Surgical Population. World Neurosurg. 2020 Dec;144:e25-e33. doi: 10.1016/j.wneu.2020.06.241. Epub 2020 Jul 9. PMID 32652276
- [Background] 5. Ito, H., Tsuchiya, J., & Asami, G. (1934). A New Radical Operation for Pott's Disease. The Journal of Bone and Joint Surgery, 16(3), 499-515.
- [Background] 6. O'Brien, M. F., Kirby, R. P., Hoyle, R. M., & Hostin, R. (2015). Anterior Access to the Thoracic and Lumbar Spine. In R. W. Hald, F. J. Schwab, C. I. Shaffrey, & J. A. Youssef, Global Spinal Alignment (pp. 499-509). St. Louis, Missouri: Quality Medical Publishing, Inc
- [Background] Phan K, Xu J, Scherman DB, Rao PJ, Mobbs RJ. Anterior Lumbar Interbody Fusion With and Without an "Access Surgeon": A Systematic Review and Meta-analysis. Spine (Phila Pa 1976). 2017 May 15;42(10):E592-E601. doi: 10.1097/BRS.0000000000001905. PMID 27669042
- [Background] 8. Condon, A. (2019, October 29). Beckers Spine Review. Retrieved from Healthgrades: https://www.beckersspine.com/spine/item/47316-healthgrades-100-best-hospitals-for-spine-surgery-in-the-us.html